CLINICAL TRIAL: NCT04295980
Title: Mechanism of Aphasia and Recovery of Language After the Injury of Geschwind's Territory: a Study Based on the Brain Network Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Jiao Yuming, Doctor, Beijing Tiantan Hospital
Other Study IDs: 81901175
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: AVM - Cerebral Arteriovenous Malformation; Language
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Geschwind's area BAVMs
  Interventions: Procedure: Surgical removal of the BAVMs
- Healthy controls

INTERVENTIONS:
Procedure: Surgical removal of the BAVMs — Resection the BAVM nidus by microsurgery.
  Groups: Geschwind's area BAVMs

SUMMARY:
At present, functional imaging studies have suggested that the Geschwind's territory (the inferior parietal lobe) is an important language area. It is the hub for semantics and phonetic language processing. However, the type and mechanism of aphasia after injury of Geschwind's territory and the subsequent recovery of language are still unclear. In our study based on brain injury model of brain arteriovenous malformation (BAVMs) resection, investigators found that the incidence of aphasia was higher after the injury of Geschwind's territory than after injury of the classical language area, and the type of aphasia was complicated, while the recovery rate of language disorder was high during follow-up. Investigators hypothesized that the type of aphasia may be associated with the type of brain connectivity damaged, and that reorganization of brain connections and brain network promote the recovery of language function. In this study, we aim to investigate the types of aphasia and their corresponding brain network changes after the resection of BAVMs located in the Geschwind's territory. Investigators will evaluate language function and collect multimodality images of the patients before resection of the lesions, as well as 7 days, 3 months and 6 months afterwards. In addition, the anatomical brain connectivity and brain network will also be analyzed. Our research will not only be a meaningful exploration for mechanisms of human language function damage and reorganization, but will also provide an important basis for the protection of brain function in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form;
2. The dominant hand is the right hand (evaluated by the Edinburgh hand scale);
3. BAVM located in the left inferior parietal lobe
4. No history of rupture and bleeding and neurosurgical treatment

Exclusion Criteria:

1. There are implants in the body (cardiac pacemaker, artificial femoral head, etc.);
2. The dominant hand is unclear;
3. Illiterate or other patients who can not cooperate well with cognitive function tests;
4. The history of bleeding in BAVM patients within one month;
5. History of neurosurgical treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study, we will recruit 40 patients with BAVMs located in Geschwind's area, and recruit 40 healthy subjects as healthy control.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain network of BAVMs in Geschwind's area | 2 years
  compare the brain network of the Geschwind's area BAVMs patients and normal controls
Brain network after injury of Geschwind's area | 2 years
  compare the preoperative and postoperative brain network of Geschwind's area BAVMs.
Brain network of the brain reorganization after surgery | 3 years
  After surgery, we compare the brain network before and after the reorganization.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China